CLINICAL TRIAL: NCT03462615
Title: Clinical Performance of the HRP2 HS-RDT for Malaria Diagnosis in Pregnant Women in Papua New Guinea
Brief Title: Clinical Performance of the Histidine Rich Protein 2 (HRP2) Highly Sensitive Rapid Diagnostic Test (HS-RDT) for Malaria Diagnosis in Pregnant Women in Papua New Guinea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Burnet Institute (Other); Papua New Guinea Institute of Medical Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: 7815-2/2
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Plasmodium Falciparum Malaria; Pregnancy Malaria; Diagnoses Disease
Keywords: malaria; pregnancy; diagnosis; rapid diagnostic test
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HS-RDT — A single finger-prick blood sample will be collected and used to test participants with the HS-RDT. The results of the results of the test will not be used for treatment purposes nor used to inform patient care.
  Other Names: ultra sensitive RDT

SUMMARY:
Malaria during pregnancy remains an important public health issue in endemic countries. Most cases of malaria in pregnant women are asymptomatic, and can contribute to adverse outcomes, such as maternal and neonatal anaemia as well as low birth weight. Infections that do not cause symptoms (sub-clinical infections) - particularly in low transmission settings -remain difficult to diagnose during pregnancy but can contribute to adverse outcomes e.g. growth restriction, premature birth, miscarriage and stillbirth.

The Bill & Melinda Gates Foundation (BMGF) has supported the development of an HRP2-based high sensitivity rapid diagnostic tests (HS-RDT) that has analytical sensitivity ten times better than current RDTs and a sensitivity near 80% when compared to the 'gold standard' of quantitative polymerase chain reaction (qPCR). In this regard, the new HS-RDT may be a promising diagnostic and screening test for subclinical malaria during pregnancy.

The overall aim is to compare the performance of novel high sensitivity rapid detection tests with conventional rapid diagnostic tests for Plasmodium falciparum malaria infection in pregnant women in Papua New Guinea

ELIGIBILITY:
Inclusion Criteria:

* All women must meet all the following inclusion criteria in order to be eligible to participate in the study:

  * Pregnant women attending first antenatal care visit at selected health facilities
  * Resident in the study area for at least 1 year prior to enrolment
  * Age ≥ 16
  * Willing to freely participate with signed informed consent (or, if illiterate, provide a thumbprint in the presence of an independent witness)
  * Willing to provide finger-prick blood sample

Exclusion Criteria:

* Women meeting any of the following exclusion criteria at screening will be excluded from study participation:

  * History of malaria or antimalarial drugs used in the last three months, as recalled or documented in health record
  * Presence of severe malaria as defined by WHO guidelines at the moment of recruitment.

Presence of symptoms and signs of other serious chronic disease such as severe anaemia, tuberculosis and/or central nervous system infections, as defined by WHO guidelines

Min Age: 16 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study will test samples from pregnant women aged 16 and older, self-presenting at health centres for antenatal care in this malaria-endemic setting
Sampling Method: Non-Probability Sample
Enrollment: 930 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  1.1 Estimates of sensitivity, specificity, negative predictive value, positive predictive value, and diagnostic odds ratio of HRP2 HS-RDT for the detection of P. falciparum during pregnancy, compared with conventional good quality RDTs, microscopy and LAMP in peripheral blood with qPCR as reference test.

IPD SHARING:
Plan to Share IPD: No